CLINICAL TRIAL: NCT06705023
Title: Adipose-derived Regenerative Cells Treatment for Congestive Heart Failure
Brief Title: Study to Assess Safety and Efficacy of Treating Symptomatic, Ischemic, Chronic Congestive Heart Failure Patients with an LVEF of ≤40% with Fresh, Uncultured, Autologous, Adipose-derived Regenerative Cells Isolated from Lipoaspirate.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ralf Rothoerl (Other)
Collaborators: National Scientific Medical Center, Kazakhstan (Other Government); Internationnal Foundation Medicine and Science (Unknown); Alliance of Cardiovascular Researchers (Other)
Responsible Party: Sponsor-Investigator, Ralf Rothoerl, coordinator, ISAR Klinikum
Organization: ISAR Klinikum (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Injury; LV Dysfunction; Coronary Artery Disease; Heart Failure
Keywords: congestive heart failure; adipose-derived regenerative cells; left ventricular ejection fraction; lipoaspirate; retrograde intra-cardiac venous injection; Cardiac Magnetic Resonance Imaging; Cardiac Computer Tomography; end systolic volume; end diastolic volume
MeSH Terms: conditions — Ventricular Dysfunction, Left; Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, controlled, multicenter, safety and efficacy study in patients with iHF comparing best available medical treatment plus a balloon-enhanced single i.cv. injection of UA-ADRCs isolated from lipoaspirate at point of care using the Transpose RT / Matrase system (InGeneron) in 24 patients, to best available medical treatment in 12 patients in the control group
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UA-ADRCs group (Experimental): Patients in the UA-ADRC (uncultured, autologous, adipose-derived regenerative cells) group will be treated as follows:
  1. Patients will have an outpatient liposuction procedure from the abdomen, bilateral flanks, and/or medial thigh (at least 100 mL of adipose tissue) to get cell product.
  2. Oral sedation and local anesthesia with tumescent solution will be used. Patients' vitals will be monitored and recorded during the procedure and in 1 to 2 hours post-procedure.
  3. Each patient in the UA-ADRC group will have cells isolated using the Transpose RT/Matrase system (InGeneron).
  4. Cell product testing will be assessed with the following acceptance criteria: total nucleated cell count is > 35 million cells, b) cell viability is > 75%. AE status will be monitored for 30 days post-liposuction procedure.
  5. The i.cv injection of UA-ADRCs will be given using an aseptic technique. This group will include 24 patients.
  Interventions: Biological: Uncultured, autologous, adipose-derived regenerative cells (UA-ADRCs)
- Control group (Active Comparator): Patients will receive continuation of their best guideline based medical treatment. This group will include 12 patients.
  Interventions: Other: Continuation of patient's best guideline based medical treatment

INTERVENTIONS:
Biological: Uncultured, autologous, adipose-derived regenerative cells (UA-ADRCs) — Intracardial venous injection of fresh, uncultured, autologous, adipose-derived regenerative cells isolated from lipoaspirate at the point of care.
  Arms: UA-ADRCs group
Other: Continuation of patient's best guideline based medical treatment — Patients will receive continuation of their best guideline based medical treatment.
  Arms: Control group

SUMMARY:
To investigate patients suffering from iHF and a LVEF of equal or less than 40% despite best medical treatment safety and efficacy of a single retrograde intra-cardiac venous (i.cv.) injection of UA-ADRCs isolated from lipoaspirate at the point of care, using the Transpose® RT / Matrase System (InGeneron, Houston, TX, USA) through an over-the- wire, small balloon catheter, advanced through the coronary si-nus and located within a coronary vein at the site of inter-est, versus patients on best medical treatment.

DETAILED DESCRIPTION:
The aim of the study is to investigate patients suffering from chronic congestive heart failure (iHF) and a left ventricular ejection fraction (LVEF) of equal or less than 40% despite best medical treatment safety and efficacy of a single retrograde intra-cardiac venous (i.cv.) injection of uncultured, autologous, adipose-derived regenerative cells (UA-ADRCs) isolated from lipoaspirate at the point of care. The cells will be isolated using the Transpose® RT / Matrase System (InGeneron, Houston, TX, USA) through an over-the-wire, small balloon catheter, advanced through the coronary sinus and located within a coronary vein at the site of interest, versus patients on best medical treatment.

This study hypothesizes that treatment of iHF with a balloon-enhanced i.cv. injection of UA-ADRCs isolated from lipoaspirate at the point of care using the Transpose RT / Matrase system (InGeneron) is safe and effective and is more effective than best medical treatment.

The primary objective of this study is to evaluate safety and efficacy of treating iHF with a single, balloon-enhanced retrograde i.cv. injection of UA-ADRCs. Efficacy will be demonstrated in a superiority study design by comparing improvement in global cardiac functional parameters demonstrated using cardiac magnetic resonance imaging (cMRI) or Cardiac CT, and by clinical endpoints after a single i.cv. injection of UA-ADRCs, to best medical treatment. Safety will be demonstrated by reporting major ad-verse cardiac events (MACE) and other adverse events.

A total of n=36 patients with iHF and a reduced LVEF (at ≤40%) will be randomly assigned to i.cv. injection of either UA-ADRCs (UA-ADRCs Group; n=24) or best medical treatment (Control Group; n=12). The enrollment will take place up to four study sites, among them the National Science Research Center of the Principal Investigator (Dr. Abay Baigenzhin) in Astana (Kazakhstan), will enroll 36 patients in the study. The study duration is the time to enroll patients in the study and will take 6 months. Individual follow-up time after the treatment is 6 months.

Follow-up schedule is as follows. Follow-up visits will take place at 1, 3, and 6 months post- treatment. Follow-up visit will include an assessment by cMRI, or cCT, physical examinations including echocardiography, patient-reported outcome questionnaires, control of medication usage, number of hospitalizations for cardiac conditions, and adverse event monitoring (including MACE). Those patients in the control group that have finished the 1, 3, and 6 month follow up visits will be offered to be treated with stem cell therapy as well. All remaining patients in both groups will be offered to participate in a subsequent registry study for 12 and 24-month follow-up vis-its, that could include physical examinations, patient-reported outcome questionnaires, medication usage, number of hospitalizations for cardiac conditions, and adverse event monitoring (including MACE) and cMRI or cCT. These long-term data would be compared to the corresponding baseline data.

The Primary Endpoint is to be cardiac function represented by left ventricular ejection fraction (LVEF) at 6 months assessed by cardiac MRI (cMRI) or cCT. Treatment success is defined as a 15% relative increase of LVEF from baseline to 6-month follow-up. Treatment success is expected in 65% of patients in the treatment group vs 10% in the control group. Secondary Endpoints will be assessed at baseline and at 6 months post-treatment and will include:

1. n-terminal pro-b-type natriuretic peptide (NT-proBNP),
2. 6-min walk test,
3. the Minnesota Living with Heart Failure Ques-tionnaire (MLHFQ) score,
4. need for hospitalization due to cardiac conditions, cardiac related death,
5. incidence of treatment-related adverse events (in-cluding MACE),
6. Only in patients with cMRI: relative amount of left ven-tricular scar tissue, left ventricular bull's eye segmental contracting areas.

This is a prospective, randomized, controlled, multicenter, safety and efficacy study in patients with iHF comparing best available medical treatment plus a balloon-enhanced single i.cv. injection of UA-ADRCs isolated from lipoaspirate at point of care using the Transpose RT / Matrase system (InGeneron) in 24 patients, to best available medical treatment in 12 patients in the control group.

Background Heart failure and myocardial infarction (MI) are consequences of ischemic heart disease (IHD) [1]. In recent years cell-based therapies have emerged as a promising strategy to re-generate ischemic myocardium [2-4]. However, the generally disappointing outcome of related clinical trials established a need for developing novel, more effective cell-based therapies for MI. In this regard, it is of note that the treatment of chronic MI (i.e., patients with a previous MI) (CMI) requires a different approach than the treatment of acute MI (AMI).

The amount of pluripotent stem cells has been reported to be significantly higher in adipose tissue than in bone marrow (5% to 10% vs. 0.1%) [12]. Fresh, uncultured, unmodified, autologous adipose-derived regenerative cells (UA-ADRCs) have the advantage over culture-expanded adipose-derived stem cells (ASCs) that UA-ADRCs allow for immediate usage at the point of care, combined with low safety concerns, since no culturing or modification is applied.

Several experimental studies in animal models have demonstrated the potential of UA-ADRCs for treating AMI [13-15], and a first clinical trial (APOLLO) showed promising preliminary results [16]. The investigators recently published results of a preclinical porcine study regarding the treatment of chronic ischemic heart failure (> 4 wk post-MI) with UA-ADRCs [28]. This study demonstrated that retrograde delivery of UA-ADRCs in a porcine model of chronic ischemic heart failure significantly improved myocardial function, increased myocardial mass, and reduced scar tissue formation. As part of this study, an evidence-based systematic review of the literature according to the PRISMA guidelines was conducted to examine preclinical studies on the treatment of iHF with stem cells [28].

Preliminary results from a study including 28 patients with chronic ischemic cardiomyopathy In one study evaluating the safety and preliminary efficacy of stromal vascular fraction ad-ministration (by a needle catheter into the myocardium) including 28 patients with chronic ischemic cardiomyopathy, the authors reported results from the six-minute walk test and LVEF at baseline and three and six months (with additional testing at 12 months if applicable) after treatment. LVEF increased from baseline to three and six months of follow-up. Results from a six-minute walk test showed a performance increase of about 80m from baseline to three, six, and twelve months of follow-up [18].

Results of our initial open-label Pilot Study in patients with inclusion and exclusion criteria comparable to the now designed randomized prospective study The pilot phase study for this randomized study was conducted in collaboration with the National Scientific Medical Center, Astana, Kazakhstan. Six patients were enrolled (five male, one female, NYHA class III, age 61.3±6.2 years) with the diagnosis of chronic ischemic heart failure and no improvement of symptoms or function after standard therapy for at least one month. All patients had documented coronary artery disease with evidence of myocardial injury and left ventricular dysfunction. Five out of six participants presented LVEF of ≤40%. All patients underwent liposuction under conscious sedation and local anesthesia. Lipoaspirate was processed according to the established InGeneron procedure to produce a cellular suspension of stromal vascular fraction including UA-ADRCs using the Transpose® RT / Matrase System (InGeneron, Houston, TX, USA). This cellular preparation was retrogradely injected via the coronary sinus into the corresponding coronary vein. The main outcome of interest was the change of LVEF (assessed by cMRI) from baseline to 3-6 months. In five of the six patients, an improvement in LVEF was observed. Further, adverse events reported were related to mild bruising/swelling/redness at the site of the liposuction in the abdominal area. There were no hospitalizations or health decline due to HF symptoms throughout the initial follow-up phase.

Rationale and Outcomes for Using UA-ADRCs

UA-ADRCs have several advantages over other types of cells used in and/or under investigation for regenerative cell therapy:

* UA-ADRCs do not share ethical concerns nor the risk of teratoma formation as reported for embryonic stem cells [19-21].
* Neither UA-ADRCs share the risk of tumorigenesis [22-24].
* Because UA-ADRCs are autologous cells which does not bear the risk of HLA mismatch [25-27].
* Adipose tissue is relatively easy to be harvested in most patients through liposuction. Furthermore, uncultured vascular-associated MSCs can represent up to 12% of the total population of SVF cells [28], whereas only 0.001%-0.1% of the total population of bone marrow nucleated cells are considered true stem cells [31, 32].
* Harvesting adipose tissue by liposuction is typically less invasive than harvesting bone marrow [31, 33, 34] with mini liposuction required.
* The use of fresh UA-ADRCs allows immediate usage at point of care [14, 41-43].
* When using UA-ADRCs during the same surgical procedure in an autologous and homologous way, they have not been considered as advanced therapy medicinal product (ATMP) by the European Medicines Agency [40].
* Recent studies indicated non-inferiority or even superiority of UA-ADRCs over ASCs in, for example, rescuing heart function after acute myocardial infarction [48], bone regeneration [50], and tendon regeneration [51] (see also [4]).

An optimal system for providing UA-ADRCs at the point of care should be capable of isolating the highest possible number of living ADRCs from the lowest possible amount of adipose tissue, in the shortest possible time, and providing the cells at the highest possible concentration in a final cell suspension. In this regard, it has been demonstrated in the literature that the Transpose RT / Matrase sys-tem (InGeneron, Houston, TX, USA) is the most efficient method with respect to the viable cell yield (i.e., the number of living cells / mL lipoaspirate).

Specifically, the investigators hypothesize that (i) a single i.cv injection of UA-ADRCs isolated with the Transpose RT / Matrase system (InGeneron) is safe and effective in the treatment of iHF, (ii) this therapy is statistically significantly more effective than just guideline based drug treatment, and (iii) i.cv injection of UA-ADRCs will possibly gain widespread acceptance, if safety and higher effectiveness than standard maximum drug therapy will be demonstrated by this and following multicenter randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria

* Have documented coronary artery disease with evidence of myocardial injury, LV dysfunction, and clinical evidence of heart failure
* Have an EF ≤40% by cardiac MRI
* Be receiving guideline-driven medical therapy for heart failure at stable and tolerated doses for ≥1 month before consent
* Be a candidate for right heart cardiac catheterization
* Have New York Heart Association class I, II, or III heart failure symptoms
* If a female of childbearing potential, be willing to use one form of birth control for the duration of the study, and undergo a pregnancy test at baseline and within 36 h before treatment

Exclusion Criteria

* Indication for standard-of-care surgery (including valve surgery, placement of LV assist device, or imminent heart transplantation), CABG procedure, and PCI. Candidates cannot be UNOS 1A or 1B, and they must have documented low probability of being transplanted.
* PCI within 3 months of randomization
* CABG within 3 months of randomization
* Valvular heart disease including mechanical or bioprosthetic heart valve, severe valvular (any valve) insufficiency/regurgitation within 12 month of consent, and aortic stenosis with valve area ≤1.5 cm2
* History of ischemic or hemorrhagic stroke within 90 d of consent
* History of an LV remodeling surgical procedure utilizing prosthetic material
* Presence of a pacemaker and ICD generator with any of the following limitations/conditions: manufactured before the year 2015
* Leads implanted <6 week before consent
* Non-transvenous epicardial or abandoned leads
* Subcutaneous ICDs
* Leadless pacemakers
* Pacemaker-dependence with an ICD (pacemaker-dependent candidates without an ICD are not excluded)
* Any other condition that, in the judgment of device-trained staff, would deem an MRI contraindicated
* A CRT device implanted within 3 months of consent
* An appropriate ICD firing or antitachycardia pacing for ventricular fibrillation or ventricular tachycardia within 30 days of consent
* Ventricular tachycardia (≥20 consecutive beats) without an ICD within 3 month of consent, or symptomatic Mobitz II or higher degree atrioventricular block without a functioning pacemaker within 3 months of consent
* Presence of LV thrombus
* Baseline eGFR <35 mL/min per 1.73 m2
* Poorly controlled blood glucose levels (HbA1c >10%)
* Hematologic abnormality evidenced by hematocrit <25%, white blood cell <2500 per μL, or platelet count <100 000 per μL
* Liver dysfunction evidenced by enzymes (AST and ALT) ˃ 3× the ULN
* Coagulopathy (INR ≥1.3) not due to a reversible cause (eg, warfarin and factor Xa inhibitors). Patients who cannot be withdrawn from anticoagulation will be excluded.
* HIV or active HBV or HCV
* Allergy to radiographic contrast material that cannot adequately be managed by premedication
* Known history of anaphylactic reaction to penicillin or streptomycin
* Received gene or cell-based therapy from any source within the previous 12 months
* History of malignancy within 3 years, excluding basal cell carcinoma or cervical carcinoma in situ which have been definitively treated
* Condition that limits expected lifespan to <1 year
* History of drug or alcohol abuse
* Chronic immunosuppressant therapy such as corticosteroids or TNF-α antagonists
* Cognitive or language barriers that prohibit obtaining informed consent or any study elements
* Pregnancy or lactation or plans to become pregnant in the next 12 months
* Conditions that, in the judgment of the Investigator or Sponsor, would impair enrollment, cell harvest, administration or follow-up

ALT indicates alanine aminotransferase; AST, aspartate aminotransferase; CABG, coronary artery bypass grafting; CRT, cardiac resynchronization therapy; EF, ejection fraction; eGFR, estimated glomerular filtration rate; HBV, hepatitis B virus; HCV, hepatitis C virus; HIV, human immunodeficiency virus; ICD, implantable cardioverter defibrillator; INR, international normalized ratio; LV, left ventricular; MRI, magnetic resonance imaging; PCI, percutaneous coronary intervention; TNF-α, tumor necrosis factor-α; ULN, upper limit of normal; UNOS, United Network for Organ Sharing; and Vo2 max, maximal oxygen consumption.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction at 6 months assessed by cardiac MRI or cCT | Baseline and at 6 month post-treatment
  Change / Increase in cardiac function (LVEF from baseline to 6 month follow-up). Treatment success is defined as ≥15% increase in LVEF assessed by cMRI or cCT if cMRI is not feasible.

SECONDARY OUTCOMES:
n-terminal pro-b-type natriuretic peptide | Baseline and at 6 month post-treatment
  Assessment of n-terminal pro-b-type natriuretic peptide in the blood samples of the patients.
6-min walk test | Baseline and at 6 month post-treatment
  A validated, sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Scar tissue assessment only in patients with cMRI | Baseline and at 6 month post-treatment
  Only in patients with cMRI: relative amount of left ventricular scar tissue, left ventricular bull's eye segmental contracting areas.
The Minnesota Living with Heart Failure Questionnaire (MLHFQ) score | Baseline and at 6 month post-treatment
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) Total score could range from 0 to 105, with higher scores indicating more significant impairment in health-related quality of lifescore will be applied to the patients.
New York Heart Association (NYHA) class | Baseline and at 6 month post-treatment
  Assessment of cardiac function according to New York Heart Association (NYHA) class.
Incidence of treatment-related adverse events (including MACE) | Baseline and at 6 month post-treatment
  Consists of the reported composite of total death; MI; stroke, hospitalization because of HF; and revascularization, including percutaneous coronary intervention, and coronary artery bypass graft.

CONTACTS AND LOCATIONS:
Overall Officials: Abay Baigenzhin, Prof Dr, Principal Investigator — National Scientific Medical Center; Ralf Rothoerl, Dr, Study Director — International Foundation of Medicine and Science
Locations (1):
- National Scientific Medical Center, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided
too early

REFERENCES:
- [Background] Anderson JL, Morrow DA. Acute Myocardial Infarction. N Engl J Med. 2017 May 25;376(21):2053-2064. doi: 10.1056/NEJMra1606915. No abstract available. PMID 28538121
- [Background] Ma T, Sun J, Zhao Z, Lei W, Chen Y, Wang X, Yang J, Shen Z. A brief review: adipose-derived stem cells and their therapeutic potential in cardiovascular diseases. Stem Cell Res Ther. 2017 Jun 5;8(1):124. doi: 10.1186/s13287-017-0585-3. PMID 28583198
- [Background] Yu H, Lu K, Zhu J, Wang J. Stem cell therapy for ischemic heart diseases. Br Med Bull. 2017 Jan 1;121(1):135-154. doi: 10.1093/bmb/ldw059. PMID 28164211
- [Background] Alt E, Pinkernell K, Scharlau M, Coleman M, Fotuhi P, Nabzdyk C, Matthias N, Gehmert S, Song YH. Effect of freshly isolated autologous tissue resident stromal cells on cardiac function and perfusion following acute myocardial infarction. Int J Cardiol. 2010 Sep 24;144(1):26-35. doi: 10.1016/j.ijcard.2009.03.124. Epub 2009 May 13. PMID 19443059
- [Background] van Dijk A, Naaijkens BA, Jurgens WJ, Nalliah K, Sairras S, van der Pijl RJ, Vo K, Vonk AB, van Rossum AC, Paulus WJ, van Milligen FJ, Niessen HW. Reduction of infarct size by intravenous injection of uncultured adipose derived stromal cells in a rat model is dependent on the time point of application. Stem Cell Res. 2011 Nov;7(3):219-29. doi: 10.1016/j.scr.2011.06.003. Epub 2011 Jun 25. PMID 21907165
- [Background] Houtgraaf JH, den Dekker WK, van Dalen BM, Springeling T, de Jong R, van Geuns RJ, Geleijnse ML, Fernandez-Aviles F, Zijlsta F, Serruys PW, Duckers HJ. First experience in humans using adipose tissue-derived regenerative cells in the treatment of patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2012 Jan 31;59(5):539-40. doi: 10.1016/j.jacc.2011.09.065. No abstract available. PMID 22281257
- [Background] Comella K, Parcero J, Bansal H, Perez J, Lopez J, Agrawal A, Ichim T. Effects of the intramyocardial implantation of stromal vascular fraction in patients with chronic ischemic cardiomyopathy. J Transl Med. 2016 Jun 2;14(1):158. doi: 10.1186/s12967-016-0918-5. PMID 27255774
- [Background] Swijnenburg RJ, Tanaka M, Vogel H, Baker J, Kofidis T, Gunawan F, Lebl DR, Caffarelli AD, de Bruin JL, Fedoseyeva EV, Robbins RC. Embryonic stem cell immunogenicity increases upon differentiation after transplantation into ischemic myocardium. Circulation. 2005 Aug 30;112(9 Suppl):I166-72. doi: 10.1161/CIRCULATIONAHA.104.525824. PMID 16159810
- [Background] Zhang Y, Wang D, Chen M, Yang B, Zhang F, Cao K. Intramyocardial transplantation of undifferentiated rat induced pluripotent stem cells causes tumorigenesis in the heart. PLoS One. 2011 Apr 28;6(4):e19012. doi: 10.1371/journal.pone.0019012. PMID 21552563
- [Background] Trounson A. Potential Pitfall of Pluripotent Stem Cells. N Engl J Med. 2017 Aug 3;377(5):490-491. doi: 10.1056/NEJMcibr1706906. No abstract available. PMID 28767348
- [Background] Fraser JK, Wulur I, Alfonso Z, Hedrick MH. Fat tissue: an underappreciated source of stem cells for biotechnology. Trends Biotechnol. 2006 Apr;24(4):150-4. doi: 10.1016/j.tibtech.2006.01.010. Epub 2006 Feb 20. PMID 16488036
- [Background] Ong WK, Sugii S. Adipose-derived stem cells: fatty potentials for therapy. Int J Biochem Cell Biol. 2013 Jun;45(6):1083-6. doi: 10.1016/j.biocel.2013.02.013. Epub 2013 Mar 1. PMID 23458962
- [Background] Klein SM, Vykoukal J, Li DP, Pan HL, Zeitler K, Alt E, Geis S, Felthaus O, Prantl L. Peripheral Motor and Sensory Nerve Conduction following Transplantation of Undifferentiated Autologous Adipose Tissue-Derived Stem Cells in a Biodegradable U.S. Food and Drug Administration-Approved Nerve Conduit. Plast Reconstr Surg. 2016 Jul;138(1):132-139. doi: 10.1097/PRS.0000000000002291. PMID 27348645
- [Background] Jiang T, Xu G, Wang Q, Yang L, Zheng L, Zhao J, Zhang X. In vitro expansion impaired the stemness of early passage mesenchymal stem cells for treatment of cartilage defects. Cell Death Dis. 2017 Jun 1;8(6):e2851. doi: 10.1038/cddis.2017.215. PMID 28569773
- [Background] Sheu JJ, Lee MS, Wallace CG, Chen KH, Sung PH, Chua S, Lee FY, Chung SY, Chen YL, Li YC, Yip HK. Therapeutic effects of adipose derived fresh stromal vascular fraction-containing stem cells versus cultured adipose derived mesenchymal stem cells on rescuing heart function in rat after acute myocardial infarction. Am J Transl Res. 2019 Jan 15;11(1):67-86. eCollection 2019. PMID 30787970
- [Background] Nyberg E, Farris A, O'Sullivan A, Rodriguez R, Grayson W. Comparison of Stromal Vascular Fraction and Passaged Adipose-Derived Stromal/Stem Cells as Point-of-Care Agents for Bone Regeneration. Tissue Eng Part A. 2019 Nov;25(21-22):1459-1469. doi: 10.1089/ten.TEA.2018.0341. Epub 2019 Jun 14. PMID 30734661
- [Background] Polly SS, Nichols AEC, Donnini E, Inman DJ, Scott TJ, Apple SM, Werre SR, Dahlgren LA. Adipose-Derived Stromal Vascular Fraction and Cultured Stromal Cells as Trophic Mediators for Tendon Healing. J Orthop Res. 2019 Jun;37(6):1429-1439. doi: 10.1002/jor.24307. Epub 2019 Apr 29. PMID 30977556